CLINICAL TRIAL: NCT01099514
Title: Phase II Study of Nilotinib in Metastatic Melanoma With KIT Aberrations
Brief Title: Study of Nilotinib in Metastatic Melanoma With KIT Aberrations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, Samsung medical center, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-02-026
Record Dates: First submitted 2010-04-06; First posted 2010-04-07 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Metastatic Melanoma With KIT Aberration
MeSH Terms: interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nilotinib (Experimental): Nilotinib 400 mg (2 capsules) PO BID q 28 days
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — D1~ Nilotinib 400 mg (2 capsules) PO BID q 28 days

SUMMARY:
Major response was observed to imatinib mesylate in KIT-mutated metastatic rectal melanoma (Hodi FS et al, J Clin Oncol 26:2046-2051, 2008). In the ASCO annual meeting in 2009ar, KIT mutations were reported to be present in 23% of acral and 15.2% of mucosal melanomas (Heinrich MC et al, J Clin Oncol 26:2008 abstr 9016). Nilotinib is a novel tyrosine kinase inhibitor (TKI) targeting KIT, PDGFR, and Bcr-Abl and inhibiting the proliferating of both imatinib-sensitive and imatinib-resistant cells in vitro. Phase I study of nilotinib alone and in combination with imatinib in patients with imatinib-resistant gastrointestinal stromal tumors (GIST) demonstrated significant activity (72% stable disease for nilotinib alone and 56% for nilotinib/imatinib combination) (Blay JY et al, J Clin Oncol 26:2008, abstr 10553).

Thus, we propose to conduct a phase II study of nilotinib in metastatic melanoma with KIT mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven melanoma with stage IV or unresectable stage III disease
2. Documented KIT aberration
3. Adequate organ function as defined by the following criteria:

   * Serum aspartate transaminase (AST); serum glutamic oxaloacetic transaminase (SGOT)) and serum alanine transaminase (ALT); serum glutamic pyruvic transaminase (SGPT)) ≤ 2.5 x local laboratory upper limit of normal (ULN), or AST and ALT less than or equal to 5 x ULN if liver function abnormalities are due to underlying malignancy
   * Total serum bilirubin ≤ 1.5 x ULN
   * Absolute neutrophil count (ANC) ≥ 1500/µL
   * Platelets ≥ 100,000/µL
   * Hemoglobin ≥ 9.0 g/dL (may be transfused or erythropoietin treated)
   * Serum calcium ≤ 12.0 mg/dL
   * Serum creatinine ≤ 1.5 x ULN
4. Patients with CNS metastasis must have stable neurologic function without evidence of CNS progression within 8 weeks
5. May have previous adjuvant therapy with interferon, vaccines or therapy with IL-2, chemotherapy
6. At least one measurable lesion by RECIST criteria
7. ECOG PS 0-2

Exclusion Criteria:

1. Major surgery or radiation therapy within 4 weeks of starting the study treatment.
2. History of or known carcinomatous meningitis, or evidence of symptomatic leptomeningeal disease on screening CT or MRI scan.
3. Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥ 2.
4. QTc > 470 msec on baseline EKG.
5. Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-08; Primary Completion 2013-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
response rate | 1~2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Cancer Center, Seoul, South Korea